CLINICAL TRIAL: NCT00585598
Title: Evaluation of Supralaryngeal Airway Removal During Initial Resuscitation of the Trauma Patient
Status: Completed | Type: Observational
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Other Study IDs: H-2006-0198
Record Dates: First submitted 2007-12-26; First posted 2008-01-03 (Estimated); Last update posted 2015-10-08 (Estimated); Status verified 2015-10

CONDITIONS: Replacement of Supralaryngeal Airway

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: all patients that are admitted to the trauma bay with a supralaryngeal airway
  Interventions: Other: replacing supralaryngeal airway with ET tube

INTERVENTIONS:
Other: replacing supralaryngeal airway with ET tube — changing tube in trauma bay

SUMMARY:
In the trauma setting, if a patient has arrived in the trauma bay with an ETC/King LT-D in place, it has traditionally been immediately exchanged out for an ETT upon arrival. The timing of the exchange has never been adequately defined in terms of safety. This study is a prospective clinical trial designed to evaluate the safety of supralaryngeal, ETC/King LT-D tube, exchange [either in the operating room (if immediate surgery is required) or after stabilization in the trauma bay/intensive care unit according to the protocol adapted previously by UWHC.

DETAILED DESCRIPTION:
The esophageal tracheal combitube (ETC) was first marketed in 1987 by Frass, Frenzer, and Zahler as an alternative airway to traditional endotracheal intubation. The combitube is a polyvinyl chloride double lumen supraglottic airway that can be placed blindly, quickly, and with minimal training. The device is available in two sizes, 37F for small adults (4-6 feet tall) and 41F for larger adults (up to 198 cm height). It is now widely used in Wisconsin for the pre-hospital airway management algorithm for trauma patients.

The combitube is designed with two lumens including a pharyngeal lumen (blind distal end and a blue proximal end which allows communication with the airway via holes positioned just above the lower pharynx) and a tracheal lumen (clear, short proximal portion and open distal portion). The device also has two balloons to allow for adequate ventilation and oxygenation while minimizing the risk of aspiration. The oropharyngeal balloon is located above the pharyngeal perforations and when inflated (85 - 100 mL of air) seals the oral and nasal cavity. The distal balloon is positioned just above the distal tracheal lumen opening and will seal either the esophagus or the trachea depending upon the positioning when inflated.

The King LT-D is designed with one lumen, two ventilation apertures located between two inflatable cuffs. The distal cuff/balloon seals the esophagus. The proximal cuff/balloon seals the oropharynx. Ventilation occurs through the proximal end of the tube.

Multiple clinical trials have been undertaken examining the safety and efficacy of the ETC & King LT-D used in the pre-hospital setting. In general, the ETC device has shown superiority to the laryngeal mask airway (LMA), oral airway/bagged mask ventilation, and the pharyngeal tracheal lumen airway in terms of success rate of insertion, ventilation, and complication rates. In-hospital use, including use in elective operative cases up to 6 hours duration and in cardiac arrest necessitating CPR, has been studied in a more limited fashion. However, small clinical trials have supported the use of ETC & King LT-D as a first line rescue airway when ETT is not possible. In addition, several studies have shown equivalence of ventilation and oxygenation between ETT and ETC used in CPR, in the operating suite, and in the ICU setting. However, most clinicians still view the supralaryngeal ETC/King LT-D as primarily rescue airways.

Although technically possible to maintain an airway with the supralaryngeal ETC/King LT-D, endotracheal intubation has been the gold standard. In the trauma setting, if a patient has arrived in the trauma bay with a supralaryngeal airway in place, it has traditionally been exchanged out for an ETT during the primary survey (initial assessment). This exchange is possible using a number of techniques widely described in the literature. Although the skilled anesthesiologists reportedly can do this exchange safely and rapidly according to a limited number of clinical trials, the safety of the exchange during the primary survey and initial resuscitation of the trauma patient has not been well documented.

This study is a prospective clinical trial designed to evaluate the exchange of the supralaryngeal airway immediately upon arrival to the trauma bay according to the UWHC previously adopted protocol.

ELIGIBILITY:
Inclusion Criteria:

* All trauma patients arriving in the trauma bay with an ETC (combitube) or King LT-D

Exclusion Criteria:

* none

Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All trauma patients arriving in the trauma bay with an ETC (combitube) or King LT-D in place will be included. The Trauma Chief resident and/or Andrea Williams, Trauma Program Specialist, will identify patients coming into the UWHC ED with supralaryngeal airways. They will concurrently or retrospectively (within 72 hours) collect data from the subjects chart or WISCR. Many of the patients arrive as unidentified persons with unknown ages. Therefore, pediatric patients will also be included. In addition, most have no consentable family readily available and the patients will not have their clinical course altered in any way by being part of this study.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2006-08; Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
efficacy of our protocol | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Lee D Faucher, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States